CLINICAL TRIAL: NCT00244816
Title: Phase II Open-Label Study of Weekly Taxoprexin® (DHA-paclitaxel) Injection as Treatment of Patients With Metastatic Uveal (Choroidal) Malignant Melanoma
Brief Title: Taxoprexin® Treatment for Advanced Eye Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01-04-22
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — docosahexaenoyl-paclitaxel; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Taxoprexin (Experimental): Taxoprexin 500 mg/m² intravenously every week
  Interventions: Drug: Taxoprexin

INTERVENTIONS:
Drug: Taxoprexin — Administered by intravenous infusion over 1 hour infusion for 5 consecutive weeks in a 6-weeks cycle.
  Other Names: Docosahexaenoic acid (DHA)-paclitaxel

SUMMARY:
To evaluate objective response rate and duration of response to weekly Taxoprexin®.

To evaluate the safety profile of weekly Taxoprexin® in this patient population.

To evaluate overall survival in the same patient population. To evaluate time to disease progression, and the time to treatment failure in patients with metastatic choroidal melanoma being treated with weekly Taxoprexin® Injection.

DETAILED DESCRIPTION:
This is a Phase II open-label study of weekly Taxoprexin® Injection in patients with metastatic choroidal melanoma who may be previously untreated or have received one prior systemic cytotoxic regimen for advanced disease. Patients may not have been treated previously with taxanes. Patients may have been previously treated with immunological agents including interleukin-2 and vaccines. Patients will receive Taxoprexin® Injection at a dose of 500mg/m2 intravenously by 1-hour infusion weekly for the first five weeks of a six week cycle. Treatment will continue until progression of disease, intolerable toxicity, refusal of continued treatment by patient or Investigator decision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic or cytologic confirmation of malignant eye melanoma, and documented metastatic disease.
2. Patients must have at least one unidimensionally measurable lesion.
3. Patients may be previously untreated or may have received one prior systemic chemotherapy regimen for metastatic disease. Patients may not have been treated previously with taxanes. Prior treatment with immunotherapy or vaccine therapy is allowed.
4. At least 6 weeks (42 days) since any prior immunotherapy, cytokine, biologic, vaccine or other therapy.
5. At least 4 weeks (28 days) since prior radiotherapy to > 20% of the bone marrow and prior adjuvant chemotherapy.
6. Lesions being used to assess disease status may not have been radiated or if so, must have progressed during or after radiation therapy.
7. Patients must have Eastern Cooperative Oncology Group performance status of 0 - 2.
8. Patients must be at least 13 years of age.
9. Patients must have adequate liver and renal function.
10. Patients must have adequate bone marrow function.
11. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution.

    -

Exclusion Criteria:

1. Patients who have received prior therapy with any taxane.
2. Patients whose site of primary melanoma is not in the choroid(eye).
3. Patients who have a past or current history of neoplasm other than the entry diagnosis, except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix or other cancers treated for cure and with a disease-free survival longer than 5 years.
4. Patients with symptomatic brain metastasis (es).
5. Patients who are pregnant or nursing and patients who are not practicing an acceptable method of birth control. Patients may not breastfeed while on this study.
6. Patients with current active infections requiring anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals).
7. Patients with current peripheral neuropathy of any etiology that is greater than grade one (1).
8. Patients with unstable or serious concurrent medical conditions are excluded.
9. Patients with a known hypersensitivity to Cremophor.
10. Patients with Gilbert's Syndrome.
11. Patients must not have had major surgery within the past 14 days.
12. Patients must not receive any concurrent chemotherapy, radiotherapy, or immunotherapy while on study.
13. Known HIV disease or infection.

    -

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved an Objective Complete Response (CR) or Partial Response (PR) | Assessed every 6 weeks, up to 24 months
  Antitumor response was defined as the percentage of participants who achieved an objective response (Confirmed Response [CR] or Partial Response [PR]), confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. Response was based on the blinded radiological review using Response Evaluation Criteria in Solid Tumors (RECIST) response guidelines, Version 1.0.
  A complete response was defined as a disappearance of all target lesions determined by 2 consecutive observations not less than 4 weeks apart.
  Partial response was defined as a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as reference the baseline sum of LD determined by 2 consecutive observations not less than 4 weeks apart.

SECONDARY OUTCOMES:
Time to Progression (TPP) | Assessed every 6 weeks until progression or death, up to 24 months
  Progression free survival time was defined as the time from the day of randomization to the start of documented progression, based on the blinded radiological review response assessment. Progressive disease was defined as a ≥ 20% increase in the sum of longest diameter (SLD) of target lesions, taking as reference the smallest SLD recorded since the treatment started or the appearance of one or more new lesions.
Time to Failure (TTF) | Baseline to stopping treatment, up to 24 months
  Time to Failure (TTF) was defined as the time from the day of randomization to the discontinuation of protocol treatment for any reason.
Overall Participant Survival | Up to 24 months
  Overall survival was defined as the time from the day of randomization to participant death or last date that participant was known to be alive, whichever occurs first. Survival data was collected every two months while participants were off-study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States